CLINICAL TRIAL: NCT07016100
Title: A Randomized Clinical Trial of Contingency Management for Gambling Disorder: Enhancing Treatment Retention and Outcomes
Brief Title: Contingency Management to Reinforce Attendance to Cognitive Behavioral Treatment for Gambling Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P24-0291
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Gambling Disorder; Gambling Problem
Keywords: contingency management
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Peer recovery specialists who facilitate recovery-related engagements will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management (Experimental): Contingency management is designed to reinforce treatment attendance. Participants will earn gift card vouchers for attendance to therapy sessions and recovery-related engagements with peer support specialists. This treatment is in addition to the standard care/ treatment as usual (cognitive behavioral therapy).
  Interventions: Behavioral: Contingency management
- Cognitive Behavioral Treatment/ Treatment as Usual (Active Comparator): This five phase cognitive behavioral therapy addresses participants' behaviors, thoughts, and emotions to help them change their gambling.
  Interventions: Behavioral: Cognitive behavioral therapy/ treatment as usual

INTERVENTIONS:
Behavioral: Contingency management — See arm description
  Arms: Contingency Management
Behavioral: Cognitive behavioral therapy/ treatment as usual — See arm description
  Arms: Cognitive Behavioral Treatment/ Treatment as Usual

SUMMARY:
The aim of this study is to conduct a trial to investigate the effectiveness of adding contingency management treatment (CM) to standard care cognitive behavioral therapy (CBT) for the treatment of gambling disorder to increase attendance to treatment. CM will be used to incentivize therapy session attendance with a therapist and engagement in recovery-related engagement with a peer recovery specialist. The proposed research will evaluate whether CM can enhance the overall effectiveness of CBT, the most widely tested treatment for individuals with gambling disorder.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) has been established as the most efficacious treatment for gambling disorder. Unfortunately, 39% of those who seek treatment dropout before completing the prescribed treatment dose, a rate that is markedly higher than found with substance use treatment (30%) and mental health treatment (20%). Increasing attendance means more time to learn the skills needed to create and sustain change and, therefore, enhance treatment outcomes. To date, there has been a dearth of research on how to keep people in CBT for gambling disorder. A logical and promising option is using contingency management (CM), where tangible incentives (i.e., vouchers) are provided upon completion of a target behavior, such as treatment attendance. CM has robust support for increasing attendance to substance use treatment (68% of participants receiving CM increase their attendance). Surprisingly, CM has not been tested to motivate attendance in gambling treatment. The current project proposes to conduct a randomized controlled trial to establish the preliminary effectiveness of CM for the treatment of gambling disorder. CM will be used to incentivize attendance to CBT therapy sessions and engagement in peer recovery specialist (PRS)-facilitated recovery support activities. PRS are individuals with lived experience with recovery who use their personal experience and training to create opportunities for tailored support as a client seeking treatment navigates recovery. The selected CM protocol will provide direct gift card payments each time the participant attends a scheduled therapy or recovery activity session. Payments will start at $30 for a therapy session and $10 for a PRS-led activity session and escalate over 8 weeks of treatment. Participants will be recruited from those seeking treatment at our well-established gambling treatment center. All participants will receive a standard course of CBT treatment that includes weekly therapy sessions and PRS-support activities. Participants will be randomized to receive either CBT treatment as usual or CM+CBT, where participants will attend treatment as usual, and each session attended will be monetarily reinforced. The investigators will explore between treatment group changes in gambling behavior, treatment engagement, and other clinical covariates in these individuals at post-treatment and at a 3-month follow-up. Treatment gains will not be limited to strictly abstinence-focused outcomes and will allow for the coding of quantitative and qualitative decreases in gambling behavior and harm, and a calculation of the percentage of individuals who meet their self-selected treatment goal (which can range from abstinence to harm reduction). Results will instrumentally further our present understanding of how to enhance motivation for treatment attendance and clarify the mechanisms of CBT for gambling disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 or older
2. Seeking treatment for gambling-related concerns at The Gambling Clinic
3. Available to meet weekly for eight treatment sessions without a known structural barrier to continuation that could interfere with study conclusions (e.g., planned relocation out of state).
4. Proficient in English (assumed by request of gambling treatment in English).
5. Must be physically present in the US.

Exclusion Criteria:

1. Minors under the age of 18.
2. Recent history of psychotic symptoms or suicidal intent
3. Not proficient in English.
4. Seeking gambling treatment for someone other than themselves (e.g., a loved one).
5. Will not be available for a full eight weeks of study participation.
6. Not physically present in the US.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of sessions attended out of total | From treatment start to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Frequency of days gambled | From 30 days prior to treatment start to the end of the 3-month follow-up window
  Number of days gambled per month
Net monetary expenditures in US $ on gambling | From 30 days prior to treatment start to the end of the 3-month follow-up window
  Money spent gambling per month
Number of gambling symptoms | From 30 days prior to treatment start to the end of the 3-month follow-up window
  Quantity of gambling disorder symptoms reported in the past month

CONTACTS AND LOCATIONS:
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States